CLINICAL TRIAL: NCT06555185
Title: Acute Responses to a Potentiation Warm-up Protocol on Sprint and Change of Direction in Female Football Players: a Randomized Controlled Study
Brief Title: Acute Responses to a Potentiation Warm-up Protocol in Female Football Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2022/03
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Athletic Performance
Keywords: performance enhancement; warm-up; sprint; change of direction; women's football

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Potentiation warm-up protocol with jumps combined with sprints with change of direction.
  Interventions: Other: Potentiation warm-up protocol
- Control group (Active Comparator): Usual warm-up exercises as previously used by the whole team.
  Interventions: Other: Usual warm-up protocol

INTERVENTIONS:
Other: Potentiation warm-up protocol — The intervention protocol consisted of i) 1st set - six hurdle jumps, with a distance of 70 cm between each, followed by a 15-m sprint with COD; (ii) 2nd set - six lateral hurdle jumps (three to the left and three to the right) followed by a 10-m sprint with COD; (iii) 3rd set - six bouncy strides, followed by a 15-m sprint with COD; (iv) 4th set - six broad jumps followed by a 10-m sprint with COD. All COD circuits had different configurations, changing the sprint distance and the angle of the COD curve. All repetitions and sets were separated by 90-second recovery intervals, and each set was performed three times.
  Arms: Experimental group
Other: Usual warm-up protocol — The usual warm-up consisted of (i) The first phase included dynamic stretching and drills to increase body temperature. This phase lasted 5-min and included slow jogging, light skipping, and dynamic stretches for hip flexors, glutes, quads, hamstrings, abductors, gastrocnemius and lower limb joints. (ii) The second phase was composed of exercises that intended to mimic specific movements of the football match, both with and without ball possession. This phase lasted 15 minutes and included exercises with and without possession of the ball, such as acceleration, COD, jumping over hurdles, and playful games with ball possession. In this group, the players only rested in a slow jog when they moved from the first to the second phase.
  Arms: Control group

SUMMARY:
This study aims to determine if the performance of female football players is affected after exposure to a potentiation protocol. It is hypothesized that performance in the selected physical tests will improve significantly and meaningfully after performing the chosen potentiation protocol compared to the control group's warm-up.

ELIGIBILITY:
Inclusion Criteria:

* players from any playing position (except goalkeepers) able to train without limitations.

Exclusion Criteria:

* players with any existing medical conditions that could compromise participation.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Agility T-test | First moment: beginning of the first training session; Second moment: at the end of the third week, after the fourth protocol session had been completed.
  Used to determine speed with directional changes such as forward sprinting, left and right side shuffling.
40-m sprint test | First moment: beginning of the first training session; Second moment: at the end of the third week, after the fourth protocol session had been completed.
  After a 5 s countdown, the participants ran forward following the route marked by cones, one at 0m indicating the start place and the other at 40m indicating the finish place. Participants started the test from a standing start position with the front foot approximately 2 cm behind the first cone.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Baptista, PhD, Study Director — Faculty of Science and Technology, UiT The Arctic University of Norway
Locations (1):
- Futebol Clube de Famalicão, Famalicão, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Raw data used for the study will be available in a public repository.
Time Frame: Raw data is already uploaded into a public repository and is intended to stay available without a date limit.
Access Criteria: No access criteria will be established.
URL: https://data.mendeley.com/datasets/2cwcz2vx4v/1

REFERENCES:
- [Derived] Zylberberg T, Martins R, Pettersen SA, Afonso J, Matias Vale Baptista IA. Acute responses to a potentiation warm-up protocol on sprint and change of direction in female football players: a randomized controlled study. BMC Sports Sci Med Rehabil. 2024 Nov 12;16(1):230. doi: 10.1186/s13102-024-01015-z. PMID 39533363
- Available data/document: Individual Participant Data Set: 10.17632/2cwcz2vx4v.1 — https://data.mendeley.com/datasets/2cwcz2vx4v/1

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT06555185/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/85/NCT06555185/ICF_001.pdf